CLINICAL TRIAL: NCT02321033
Title: Einfluss Der Postprandialen Glykämie Auf Inaktivitäts-induzierte Veränderungen im Stoffwechsel
Brief Title: Influence of Daylong Glycemia on Detraining Induced Metabolic Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Lazysportsmen2014
Record Dates: First submitted 2014-08-21; First posted 2014-12-22 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: glycemic index; inactivity; insulin sensitivity; metabolic flexibility; arterial stiffness; young men
MeSH Terms: conditions — Sedentary Behavior; Insulin Resistance | interventions — Carbonated Beverages

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- low glycemic index (Experimental): palatinose in soft drinks
  Interventions: Dietary Supplement: soft drinks
- high glycemic index (Experimental): sucrose plus maltodextrin in soft drinks
  Interventions: Dietary Supplement: soft drinks

INTERVENTIONS:
Dietary Supplement: soft drinks — soft drinks with palatinose and maltodextrin

SUMMARY:
Aim of the study is to investigate the impact of glycemic index (provided as soft drinks) on changes in insulin sensitivity, metabolic flexibility, and arterial stiffness in response to detraining.

The investigators hypothesize that low glycemic soft drinks decrease the detraining-induced impairment of insulin sensitivity, metabolic flexibility and arterial stiffness.

DETAILED DESCRIPTION:
The duration of the study is 7 weeks: two x 2 weeks intervention (phase A and phase B) with 3 weeks washout phase inbetween. Each 2-week intervention phase consists of an active week followed by an inactive week.

in phase A subjects consume high GI (maltodextrin and sucrose) soft drinks during the inactive week. In phase B subjects consume a low GI soft drink (palatinose) during the inactive week.

subjects were randomly assigned to either start with phase A or with phase B (cross over design).

During the whole study duration all food is provided (55% CHO, 30% fat, 15% protein)

Physical activity will be assessed by a step counter (active phase 7000-10000 steps/d and inactive phase 3000-4000 steps/d).

ELIGIBILITY:
Inclusion Criteria:

* normal weight men,
* age 18-35 y,
* active life style,
* > 300 min sports/week

Exclusion Criteria:

* food allergies,
* regular use of medication,
* smoking,
* chronic disease,
* vegan/vegetarian diet

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Influence of GI on inactivity-induced changes in insulin sensitivity as measured by an OGTT | the difference between the end of each 1 week activity phase (day 7 vs. day 14, low vs. high physical activity) is compared between high GI and low GI intervention
  Influence of GI (glycemic index) on detraining-induced changes (difference between the end of high activity and low activity phases) in insulin sensitivity Insulin sensitivity is assessed by HOMA and Matsuda indices

SECONDARY OUTCOMES:
Influence of GI on inactivity-induced changes in metabolic flexibility as measured by indirect calorimetry (RER, respiratory exchange ratio) | the difference between the end of each 1 week activity phase (day 7 vs. day 14) is compared between high GI and low GI intervention
  Impact of GI on inactivity induced changes in metabolic flexibility Metabolic flexibility is defined as the body´s ability to adapt fuel oxidation to changing fuel availability and energy demand It is measured as change in fasting RER (fasting metabolic flexibility) and change in RQ (difference between the end of high activity and low activity phases) after an oral glucose tolerance test (postprandial metabolic flexibility)

OTHER OUTCOMES:
Influence of GI on inactivity-induced changes in parameters of arterial stiffness as measured by pulse wave velocity | the difference between the end of each 1 week activity phase (day 7 vs. day 14) is compared between high GI and low GI intervention
  impact of GI on inactivity-induced changes (difference between the end of high activity and low activity phases) in arterial stiffness (as assessed by pulse wave velocity)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bosy-Westphal, Prof PhD, Principal Investigator — University of Hohenheim, Stuttgart, Germany
Locations (1):
- Institute of Nutritional Medicine, University of Hohenheim, Stuttgart, Germany